CLINICAL TRIAL: NCT04210024
Title: Social Network Analysis to Identify Community Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brittany L Smalls (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Brittany L Smalls, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 45657; 1K01DK116923 (NIH)
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Type2 Diabetes
Keywords: Diabetes Empowerment Education Program (DEEP); social network analysis; Integrated Behavioral Model (IBM); rural; community; Appalachia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rural-Dwelling Community Members/Residents (Other): Rural-dwelling adults will be interviewed to map their social network structure, determine the types of social support provided by members of their social network, and identify key players within these networks. A subset of participants (~4) will be identified as Community Health Workers and will receive training with the Diabetes Empowerment Education Program (DEEP).
  Interventions: Other: Diabetes Empowerment Education Program

INTERVENTIONS:
Other: Diabetes Empowerment Education Program — Individuals identified as Community Health Workers will participate in the Diabetes Empowerment Education Program (DEEP™). DEEP, is an education curriculum designed to help people with pre-diabetes, diabetes, relatives and caregivers gain a better understanding of diabetes self-care. Classes last a total of six weeks, providing participants with eight unique learning modules. Health literacy will be assessed before and after participating in DEEP.

SUMMARY:
The objective of this study is to recruit influential community members using Snowball Sampling Methods. Community members identified through social network analysis as influential and well-connected will be trained as community health workers (CHW) using the Diabetes Empowerment Education Program (DEEP). These CHW will be used in a future trial to educate other members of the community.

DETAILED DESCRIPTION:
The proposed research employs the Integrated Behavior Model (IBM) to address fundamental drivers of behavior for older rural-dwelling adults with type-two diabetes mellitus (T2DM) in the context of their social network. Social network analysis (SNA) is characterized as the examination and interpretation of relational connections. This approach can be used to map social networks and understand relationships between individuals as it pertains to social support. Snowball recruitment methods will be used to recruit participants in this study. In Aim 1, individuals who are connected to several individuals within their community and have the capacity to influence norms that hinder T2DM self-care will be identified. Ten individuals who have received medical care from the Center of Excellence in Rural Health (CERH) within the past 12 months will be identified. Initial recruitment will be conducted by a community liaison in Leslie County. This core group of 10 "seeds" will be used to conduct the first wave of interviews. Since the aim of social network analysis is to understand a community by mapping the relationships that connect them as a network, each seed will be asked to identify 3 persons believed to be influential in their community. Those who are identified in wave 1 will also be asked to identify 3 people each from their community who are also respected as leaders and can be trusted to provide health-related information to community members. This process will continue for 4 waves of recruitment (N˜200).

Participants will be asked to provide demographic information including age, sex, race/ethnicity, education, employment status, contact information (address, telephone number, email). An interview guide will be adapted from a previously published intervention assessing social networks and health behavior informed by preliminary data and the expert opinion of my team of mentors and collaborators. The interviews will begin with two broad general questions asking "who" is included in their social network and "how" members of the social network provide social support; using open-ended questions to elicit maximal information with minimal bias. Interview questions will explore the following domains: size and structure of social network; resources available through social network; beliefs of those in social network regarding general healthy behavior; knowledge of available healthy lifestyle choices; and perceived acceptable healthy behaviors (social norms). Data will be collected from CHWs pre- and post-training to assess the following: T2DM knowledge: Diabetes Knowledge Questionnaire (DKQ) a 24-item survey that has a reliability coefficient of 0.78 and showed sensitivity to a T2DM knowledge intervention. Health literacy: Newest Vital Sign (NVS) is a 6-item survey to assess health literacy comprehension and numeracy. Means and paired t-tests will be conducted to determine if health literacy and T2DM knowledge improved in each CHW during the DEEP training.

ELIGIBILITY:
Inclusion Criteria:

* residents of Leslie County, Kentucky
* speak and understand English

Exclusion Criteria:

* under 18 years of age
* unable to speak and understand English
* unable to consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Smalls, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Center for Excellence in Rural Health, Kentucky Homeplace, Hyden, Kentucky
  - Stinnett Area Community Center, Stinnett, Kentucky

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to covid, the study was paused by the institutions for 18 months. In order to get back on track with the intervention, we could not identify and train community health workers to participate in the study based on the data collected for social network analysis. Alternatively, the research coordinator administered the intervention. There were no community health works.
Groups:
- Rural-Dwelling Community Members/Residents: Rural-dwelling adults will be interviewed to map their social network structure, determine the types of social support provided by members of their social network, and identify key players within these networks. A subset of participants (~4) will be identified as Community Health Workers and will receive training with the Diabetes Empowerment Education Program (DEEP).
  This was a cohort study/community assessment and there were no study arms.
  Diabetes Empowerment Education Program: Individuals identified as Community Health Workers will participate in the Diabetes Empowerment Education Program (DEEP™). DEEP, is an education curriculum designed to help people with pre-diabetes, diabetes, relatives and caregivers gain a better understanding of diabetes self-care. Classes last a total of six weeks, providing participants with eight unique learning modules. Health literacy will be assessed before and after participating in DEEP.
Period: Overall Study
Arm/Group | Rural-Dwelling Community Members/Residents
Started | 91
Completed | 91
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rural-Dwelling Community Members/Residents
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age for one participant was missing
  years
    number analyzed (Participants) | 90
    (all) | 45.54 (15.81)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant did not report this demographic
  Participants
    number analyzed (Participants) | 90
    Female | 60
    Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 91
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 91
Education [Count of Participants; unit: Participants]
  Year 12 or equivalent | 41
  Diploma or Advanced Diploma | 17
  Bachelor Degree | 13
  Graduate certificate/diploma | 2
  Master's Degree | 4
  None of the above | 14
Employment Status [Count of Participants; unit: Participants]
  Employed Full-time | 35
  Employed Part-time | 10
  Retired | 7
  Unable to work/Disabled | 17
  Unemployed | 22
Insurance [Count of Participants; unit: Participants]
  None | 3
  Private | 27
  Medicare | 16
  Medicaid | 29
  Military Care | 1
  Other Insurance | 15
Difficulty understanding or speaking English [Count of Participants; unit: Participants]
  Never | 86
  Rarely | 1
  Sometimes | 2
  Often | 0
  Always | 1
  Don't Know | 1
Reading or writing English [Count of Participants; unit: Participants]
  Never | 78
  Rarely | 5
  Sometimes | 5
  Often | 1
  Always | 1
  Don't know | 1
Marital Status [Count of Participants; unit: Participants] — Population: 1 participant did not report this demographic
  Participants
    number analyzed (Participants) | 90
    Married | 23
    Separated/Divorced | 29
    Widowed | 8
    Never Married | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Diabetes Knowledge
Description: The change in participants' knowledge of Type 2 Diabetes Mellitus (T2DM) will be assessed using the Diabetes Knowledge Questionnaire (DKQ) pre- and post-training with the DEEP program. The DKQ is a 24-item survey assessing diabetes knowledge. Scores range from 0-24; higher scores indicate increased knowledge of diabetes.
Time Frame: 6 weeks
Population: Data not collected for this outcome
Arm/Group | Rural-Dwelling Community Members/Residents
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Health Literacy
Description: Change in health literacy pre- and post-education with the DEEP program will be assessed using the Newest Vital Sign (NVS) survey tool. NVS assesses health literacy based on participant interpretation of food labels. Scores range from 0-6. Lower scores indicate a high likelihood of limited literacy while higher scores indicate adequate literacy.
Time Frame: 6 weeks
Population: Data not collected for this outcome
Arm/Group | Rural-Dwelling Community Members/Residents
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: No adverse event data to report
Arm/Group | Rural-Dwelling Community Members/Residents
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT04210024/Prot_001.pdf
  • Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04210024/ICF_000.pdf